CLINICAL TRIAL: NCT05444894
Title: A Multicenter Study to Evaluate the Safety, Tolerability, and Efficacy of a Single Dose of Autologous Clustered Regularly Interspaced Short Palindromic Repeats Gene-edited Cluster of Differentiation 34 (CD34+) Human Hematopoietic Stem and Progenitor Cells (HSPC) (EDIT-301) in Transfusion-Dependent Beta Thalassemia (TDT)
Brief Title: EDIT-301 for Autologous Hematopoietic Stem Cell Transplant (HSCT) in Participants With Transfusion-Dependent Beta Thalassemia (TDT)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Editas Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-301-BThal-001
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Transfusion Dependent Beta Thalassemia; Hemoglobinopathies; Thalassemia Major; Thalassemia Intermedia
Keywords: Beta-Thalassemia; Hemoglobinopathies; CRISPR-Cas 12a; Autologous CD34+
MeSH Terms: conditions — Hemoglobinopathies; beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EDIT-301 (Experimental): EDIT-301 (autologous gene edited (CD)34+ hematopoietic stem cells) will be administered as a one-time intravenous infusion.
  Interventions: Genetic: EDIT-301

INTERVENTIONS:
Genetic: EDIT-301 — Administered by intravenous infusion after myeloablative conditioning with busulfan.
  Other Names: renizgamglogene autogedtemcel; reni-cel

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of treatment with EDIT-301 in adult participants with Transfusion Dependent beta Thalassemia

DETAILED DESCRIPTION:
This is a Phase 1/2 single-arm, open-label, multicenter study evaluating the safety, tolerability, and efficacy of a single unit dose of EDIT-301 for autologous hematopoietic stem cell transplant in adult participants with TDT, age 18 to 35 years, inclusive

ELIGIBILITY:
Key Inclusion Criteria:

Diagnosis of Transfusion Dependent B-Thalassemia as defined by:

* Documented homozygous β-thalassemia or compound heterozygous β-thalassemia including β-thalassemia/hemoglobin E (HbE) based on historical data in medical records, and
* History of at least 100 mL/kg/year or 10 U/year of packed red blood cell (RBC) transfusions in the 2 years prior to signing informed consent
* Clinically stable and eligible to undergo autologous HSCT
* Karnofsky Performance Status ≥ 70

Key Exclusion Criteria:

* Available 10/10 human leukocyte antigen (HLA)-matched related donor
* Prior HSCT or contraindications to autologous HSCT
* Participants with associated a history of α-thalassemia and > 1 alpha chain deletion, or alpha multiplications as documented in medical records
* Participants with a history of other inherited hemoglobinopathy or thalassemic mutation (Hb S, C, D or other) as documented in medical records
* Prior receipt of gene therapy
* Inadequate bone marrow function, as defined by white blood cell count of < 3 x 10^9/L or a platelet count < 100 x 10^9/L (without hypersplenism), per investigator judgement
* Inadequate organ function
* Advanced liver disease
* Any prior or current malignancy, or immunodeficiency disorder,
* Immediate family member with a known or suspected Familial Cancer Syndrome
* Clinically significant and active bacterial, viral, fungal, or parasitic infection

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving engraftment defined as neutrophil engraftment (defined as demonstrating absolute neutrophil count (ANC) ≥ 0.5 x 10^9/L post EDIT-301 infusion for 3 consecutive measurements obtained on different days) | EDIT-301 infusion (Day 0) to 42 days post EDIT-301 infusion
Frequency and severity of adverse events (AEs) (incidence of AEs and Grade 3 or higher serious adverse events, using National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v.5.0) | Screening through up to 24 months post EDIT-301 infusion

SECONDARY OUTCOMES:
Kinetics of HSPC engraftment | EDIT-301 infusion (Day 0) to first day in which 3 consecutive measurements obtained on different days demonstrate ANC ≥ 0.5 x 10^9/L up to 24 months post EDIT-301 infusion
  Time to neutrophil engraftment
Kinetics of HSPC engraftment | EDIT-301 infusion (Day 0) to first day of 3 consecutive measurements of platelets ≥ 50 x 10^9/L for at least 1 week following the last platelet transfusion and 10 days following thrombopoietin mimetics use up to 24 months post EDIT-301 infusion.
  Time to platelet engraftment
Incidence of transplant related mortality | EDIT-301 infusion (Day 0) through Day 100 post EDIT-301 infusion and from EDIT-301 infusion (Day 0) through 12 months post EDIT-301 infusion
Incidence of all-cause mortality | Screening through up to 24 months post EDIT-301 infusion
Proportion of alleles per participant with intended genetic modification present in peripheral blood over time | EDIT-301 infusion (Day 0) through up to 24 months post EDIT-301 infusion
Proportion of alleles per participant with intended genetic modification present in bone marrow cells over time | EDIT-301 infusion (Day 0) through up to 24 months post EDIT-301 infusion
Change in the fetal hemoglobin (HbF) concentration compared to baseline overtime | Baseline through up to 24 months post EDIT-301 infusion
Change in the total hemoglobin concentration compared to baseline overtime | Baseline through up to 24 months post EDIT-301 infusion
Proportion of participants with hemoglobin concentration ≥ 9 g/dL | EDIT-301 infusion (Day 0) through 3, 6, 12 months up to 24 months post EDIT-301 infusion
Proportion of participants achieving the sustained transfusion reduction (TR) for at least 6 months and at least 12 months from 3 months post-EDIT-301 infusion | 3 months post EDIT-301 infusion through up to 24 months post EDIT-301 infusion
Proportion of participants achieving the sustained transfusion independence (TI) for at least 6 months and, at least 12 months from 3 months post EDIT-301 infusion | 3 months through up to 24 months post EDIT-301 infusion
Change in parameters of iron overload compared to baseline over time | Baseline through up to 24 months post EDIT-301 infusion
Proportion of participants receiving iron chelation therapy over time | EDIT-301 infusion (Day 0) through up to 24 months post EDIT-301 infusion

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - University of California San Francisco, Oakland, California
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center - Department of Pediatrics, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Tristar Medical Group Children's Specialists/Sarah Cannon Center for Blood Cancers, Nashville, Tennessee
- Princess Margaret Cancer Centre-University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No